CLINICAL TRIAL: NCT05555134
Title: INHALATION CHAMBER MANAGEMENT IN PEDIATRICS: EFFICACY OF AN EDUCATIONAL INTERVENTION IN PATIENTS DIAGNOSED WITH BRONCHOSPASM AND THEIR FAMILY CAREGIVERS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Belén de la Rosa, Belén de la Rosa Roch, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PuertadeHierro.
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Bronchospasm
MeSH Terms: conditions — Bronchial Spasm | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): receive usual care
- EXPERIMENTAL (Experimental): receive the educational intervention, along with usual care
  Interventions: Behavioral: educational intervention

INTERVENTIONS:
Behavioral: educational intervention — will also have an extra educational intervention, a group intervention (4-6 people) through a one-hour training session via zoom, which will be given by the PI (extensive experience in the subject) a week after discharge from the ER. Information will be reinforced and doubts will be solved
  Arms: EXPERIMENTAL

SUMMARY:
Several studies show that unnecessary and frequent visits to the emergency department for bronchospasm care are associated with inadequate management of inhalers and poor education on the approach to respiratory distress. Main objective: To determine the degree of frequentation to the pediatric emergency department for bronchospasm at 1, 3 and 6 months after the educational intervention. Design: Randomized controlled clinical trial with two groups: EXPERIMENTAL will receive the educational intervention, along with usual care, and CONTROL will receive usual care. Subjects: pediatric patients (2-15 years) diagnosed with bronchospasm; in home treatment with inhalation chambers; and their parents. Emergency Department recruitment. Follow-up at home

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2-15 years of age attending the Pediatric Emergency Department of the Hospital Universitario Puerta de Hierro Majadahonda (HUPHM) with a mild, moderate or severe bronchospasm crisis and who have used the inhalation chambers on at least one occasion; with autonomy in the use of the inhalation chambers at home

Exclusion Criteria:

* Not understanding Spanish

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
degree of frequentation to the emergency department | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Belén de la Rosa, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No